CLINICAL TRIAL: NCT06204328
Title: The Prevalence of Caregiving Burden With Influencing Factors and Effect of mHealth Psychoeducational and Benson Relaxation Technique Among Female Informal Caregivers of Cancer Patients in Bangladesh
Brief Title: Combined Effects of mHealth Psychoeducational and Benson Relaxation Technique Among Female Informal Caregivers of Cancer Patients in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, MD MARUFUR ROSHID, Principal Investigator, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NUB/ DPH/EC 2023/ 26
Record Dates: First submitted 2023-12-28; First posted 2024-01-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Caregiver Burden
Keywords: Cancer; Caregiver; Care Burden; mHealth Psychoeducation; Benson Relaxation Technique; Bangladesh
MeSH Terms: conditions — Caregiver Burden; Neoplasms

STUDY DESIGN:
Masking Description: The computer-generated simple random sampling technique will be used to select the caregiving burden of study participants for both the intervention and control groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benson relaxation technique and mHealth psychoeducation (Active Comparator): Intervention Group will receive 6 months mHealth psychoeducation & Benson Relaxation Technique
  Interventions: Other: Benson relaxation technique and mHealth psychoeducation
- Usual care (No Intervention): The usual care group will follow established and common practices by healthcare providers in these settings.

INTERVENTIONS:
Other: Benson relaxation technique and mHealth psychoeducation — Benson relaxation technique & mHealth psychoeducation (combined intervention) will receive: 6 months.
  Benson relaxation technique: Definition, benefits, and instruction about the Benson relaxation technique will be provided through recorded video, and a nurse will guide individuals face-to-face after receiving training from a physiotherapist.
  mHealth psychoeducation: There will be six sessions in a total of six months of intervention, and every session will be conducted at the beginning of each month. During each session, recorded videos based on the self-determination theory (symptom management, maintaining and enhancing relationships, problem-solving, stress and coping, self-care, and effective communication) will be provided face-to-face to the intervention group via smartphones, tablets, or handheld computers. As well as phone calls and SMS reminders will continue every week for follow-up and question and answer sessions.
  Arms: Benson relaxation technique and mHealth psychoeducation

SUMMARY:
Background: Cancer is a global health concern that places a substantial burden not only on patients but also on their informal caregivers, often family members or close friends without formal medical training. Numerous studies show that caregivers face significant burdens, which impact their physical, social, and psychological well-being. Female caregivers, often subjected to cultural expectations, face heightened challenges, contributing to higher levels of burden and emotional distress. However, the combined effectiveness of Benson relaxation techniques and mHealth psychoeducational interventions on female informal caregivers of cancer patients remains relatively unexplored.

Objective: This study aims to investigate the combined effectiveness of the mHealth psychoeducational intervention and Benson relaxation techniques to reducing caregiving burden as well as anxiety and depression, and to assess the impact on the quality of life among female informal caregivers of cancer patients in Bangladesh.

Methods: A randomized control trial study will be conducted at the Khwaja Yunus Ali Medical College and Hospital in Enayetpur, Sirajganj, Bangladesh. Computer-generated simple random sampling technique will be used to select study participants. The study period will be from April 2024 to September 2024. Data will be collected through face-to-face interviews, employing validated tools such as Zarit Burden Interview, Hospital Anxiety Depression Scale, and Bangla WHOQOL-BREF.

The intervention group will receive a combined intervention using self-determination theory (symptom management, maintaining and enhancing relationships, problem-solving, stress and coping, self-care, and effective communication) and Benson relaxation techniques through recorded videos, phone calls, and SMS reminders over six months. The control group will receive only usual care.

The study ensures ethical practices, obtains informed consent, and prioritizes data safety and confidentiality. Results will be analyzed using statistical methods, which will provide valuable information for healthcare professionals, policymakers, and researchers in the field of cancer caregiving.

DETAILED DESCRIPTION:
Chronic and non-communicable diseases represent major challenges of the twenty-first century, leading to severe consequences and societal issues for patients and communities across the globe. Cancer is a significant public health concern worldwide. Each year, cancer claims the lives of over 50 million people globally, with a particularly significant observation that 80% of these deaths occur in low- and middle-income countries. Cancer is impacting not only the patients but also their families and caregivers. Informal caregivers, who are often family members or close friends, play a crucial role in providing support and assistance to cancer patients. These caregivers usually have no knowledgeable medical training. The role of these caregivers is crucial throughout the entire disease trajectory of cancer patients, starting from the moment of diagnosis until the end stages of the illness. In the context of cancer, caregivers often face significant challenges related to the patient's treatment, symptom management, and fulfilling daily care needs. Caring for cancer patients can result in increased levels of caregiving burden, anxiety, depression, and reduced quality of life, which they encounter throughout their caregiving journey.

The prevalence of caregiving burden among caregivers of cancer patients is significant and well-established. A study published in India reported that 92.5% of caregivers experienced mild to severe levels of burden. Furthermore, a systematic review published in Cancer Nursing indicated that between 37% and 100% of family caregivers reported feeling a certain level of caregiver burden in various studies. Caregiving burden is negatively correlated with depression and anxiety. A systematic review highlighted that among the population of cancer caregivers, the prevalence of depression and anxiety was found to be 42% and 47%, respectively. This study indicated that nearly half of the caregivers experienced severe levels of depression (46%) and anxiety (53%). In addition, the demands of caregiving can result in physical, emotional, and social limitations, leading to a reduced overall quality of life. Previous studies reported that the burden of caregiving has a negative impact on the quality of life among caregivers of cancer patients. In Iran, another study discovered that as the quality of life among caregivers increased, there was a corresponding decrease in caregiver burden.

Over the past few years, there has been a growing interest in utilizing digital health technology, particularly mobile health (mHealth). As defined by the World Health Organization, "mHealth is a term used for medical and public health practice supported by mobile devices, such as mobile phones, patient monitoring devices, Personal Digital Assistants (PDAs), and other wireless devices". The mHealth involves various communication channels such as short messaging service (SMS), phone calls, online platforms, social networks, and emails to provide interventions. mHealth psychoeducational interventions can provide caregivers with accessible information, self-care tools, and resources specific to their caregiving journey which can improve their knowledge, skills, and self-efficacy, ultimately enhancing their capacity to manage caregiving responsibilities and their own well-being. A previous study published in the JMIR Mental Health journal showed the effectiveness of mHealth psychological interventions as a viable treatment approach for caregivers who experience high levels of stress or burden. In parallel, relaxation techniques are one of the non-pharmacological methods used to relieve mental health problems in various patients and their caregivers. Various relaxation techniques exist, and among them Benson's relaxation technique (BRT) is considered one of the most effective, low-cost, and straightforward methods of intervention. These techniques include mindfulness exercises that specifically treat a variety of mental and emotional symptoms, such as burden, anxiety, pain, depression, mood swings, and self-esteem problems. Previous studies have demonstrated the effectiveness of the BRT in reducing caregiving burden, anxiety and depression among various populations, including caregivers.

In Bangladesh, 1.3-1.5 million cancer patients which is added 0.2 million every year. Female caregivers play a vital role in providing personal support to patients. As a cultural expectation, women are generally expected to perform caregiving activities while also maintaining household responsibilities and familial commitments, which places an additional burden on them. Females in Bangladesh experience the most disadvantage and vulnerability for a multitude of reasons. Research has shown that female caregivers experience higher levels of burden and emotional distress than male caregivers, which has a substantial influence on life quality. However, the unique cultural context, gender inequalities, and social norms of Bangladesh might provide additional difficulties for these caregivers. It is essential to create effective interventions and support systems to alleviate their burden and improve their mental health and overall quality of life. To our knowledge, there is a significant knowledge gap, while there is growing evidence supporting the effectiveness of BRT and mHealth psychoeducational interventions separately, their combined impact on female informal caregivers of cancer patients remains relatively unexplored. This research protocol outlines a randomized controlled trial aimed at evaluating the effectiveness of combining the mHealth psychoeducational intervention and BRT in reducing these negative effects.

The results of this study are expected that the combination of mHealth psychoeducational and BRT will be effective in reducing caregiver burden, increasing psychological well-being, and improving overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Who is facing caregiving burden in the baseline screening of the study.
* Female being 18 years of age or older.
* At least 6 months of providing care to a cancer-diagnosed patient.

Exclusion Criteria:

* Refusal to collaborate with ongoing study.
* Caregivers who receive financial compensation or are employed as formal caregivers.
* Extremely traumatic events that occur during the study (such as the death of loved ones or patients, separations, etc.) or caregivers undergoing treatment with psychotropic drugs will not be included in the study.
* Without smart mobile devices at home.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Changes the caregiving burden among female informal caregivers of cancer patients in Bangladesh. | Baseline, 3 months (midline), and 6 months (endline) of intervention
  The primary outcome will be evaluated by the Zarit Burden Interview scale.
  The Zarit Burden Interview scale consists of 22 items, and each item has a 5-point Likert scale ranging from 0 to 4, whereas higher scores represent higher burden.

SECONDARY OUTCOMES:
Changes in caregivers' anxiety and depression of cancer patients. | Baseline, 3 months (midline), and 6 months (endline) of intervention
  Evaluate by using the Hospital Anxiety and Depression Scale.
  The Hospital Anxiety and Depression Scale comprises 14 items, divided into 7 questions for anxiety and another 7 questions for depression. Each item has a 4-point Likert scale, with a minimum value of 0 and a maximum value of 3. The higher score indicates high anxiety or depression.
Measuring the changes in quality of life among caregivers of patients with cancer. | Baseline, 3 months (midline), and 6 months (endline) of intervention
  Evaluate by using World Health Organization Quality of Life: Brief Version Instrument
  The World Health Organization Quality of Life Brief Version comprises 26 items rated on a 5-point Likert scale ranging from 1 to 5, with a lower score representing the least favorable outcome and a higher score representing the most favorable outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Khwaja Yunus Ali Medical College Hospital, Sirajganj, Rajshahi Division, Bangladesh

IPD SHARING:
Plan to Share IPD: No
When the data will be available and we will share the data according to the recommendations of the clinical trial registration and the requests of the journals.